CLINICAL TRIAL: NCT07256704
Title: Hypnosis and Attention in Patients With a Neurological Disease
Brief Title: Hypnosis and Attention in Patients With a Neurological Disease (Stroke, Traumatic Brain Injury and Multiple Sclerosis)
Acronym: HYPNOVA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-01374
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Stroke; Traumatic Brain Injury; Multiple Sclerosis
Keywords: Hypnosis; Attention deficit; Neurorehabilitation; Electroencephalography (EEG)
MeSH Terms: conditions — Stroke; Brain Injuries, Traumatic; Multiple Sclerosis; Attention Deficit Disorder with Hyperactivity | interventions — Hypnosis

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two groups: the hypnosis intervention group or the sham hypnosis control group.
  Arm 1: Hypnosis Intervention
  Description: Participants receive hypnosis sessions designed to improve attention and reduce fatigue.
  Arm 2: Sham Hypnosis Control
  Description: Participants receive sham hypnosis sessions serving as a control condition.
Who Masked: Participant, Outcomes Assessor
Masking Description: This study is a double-blind design, where both participants and outcome assessors are blinded to the intervention assignment. Participants will not know whether they are receiving hypnosis or sham hypnosis, minimizing expectancy and placebo effects. Outcome assessors who conduct attentional testing will also be blinded to group allocation to reduce assessment bias. Due to the nature of the intervention, the practitioner administering the sessions may be aware of the condition but will have no role in outcome assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Hypnosis Intervention
  Participants receive hypnosis sessions designed to improve attention and reduce fatigue.
  Interventions: Other: Hypnosis
- Control (Sham Comparator): Sham Hypnosis Control
  Participants receive sham hypnosis sessions serving as a control condition.
  Interventions: Other: Hypnosis

INTERVENTIONS:
Other: Hypnosis — Hypnosis sessions designed to improve attentional control and reduce fatigue in patients with neurological conditions (stroke, TBI, MS). The intervention involves guided hypnotic induction and suggestions tailored to enhance cognitive focus and energy management.

SUMMARY:
This feasibility study investigates the potential of hypnosis as a complementary therapy to improve attentional deficits and fatigue in patients with neurological diseases such as stroke, traumatic brain injury (TBI), and multiple sclerosis (MS). These patients often experience reduced spontaneous visual exploration and impaired functional independence despite current rehabilitation methods. By integrating hypnosis with standard care, and using EEG to monitor brain activity during hypnosis and sham-hypnosis sessions, this trial aims to evaluate the practicality, acceptability, and preliminary efficacy of hypnosis in enhancing attention and reducing fatigue.

DETAILED DESCRIPTION:
Neurological conditions such as stroke, traumatic brain injury (TBI), and multiple sclerosis (MS) frequently cause significant impairments in attentional abilities. Commonly accompanying symptoms include visual spatial neglect (VSN) and fatigue syndrome, which exacerbate attentional deficits. These impairments manifest notably as a reduction in spontaneous or free visual exploration (FVE), limiting patients' ability to actively scan and engage with their environment. This diminished visual exploration negatively impacts their capacity to navigate daily surroundings, compromising functional independence and overall quality of life (Chiaravalloti & DeLuca, 2008; Dillon et al., 2022; Huang et al., 2022).

Current therapeutic approaches include cognitive rehabilitation, visual exploration training, and non-invasive brain stimulation to promote neuroplasticity and functional recovery (Alashram AR, 2024; Liu-Ambrose et al., 2022; Rayegani et al., 2024; Bode et al., 2023; Lefaucheur et al., 2020). Additionally, management of fatigue focuses on energy regulation strategies in everyday life (Hersche et al., 2019). Despite these interventions, many patients continue to experience persistent attentional deficits and fatigue after rehabilitation, limiting their ability to perform daily activities and return to previous roles.

Hypnosis is emerging as a promising adjunct therapy in neurological rehabilitation. Widely used in medical fields such as pain management and mental health, hypnosis leverages the brain's ability to enter a state of focused attention and heightened cognitive receptivity, facilitating symptom relief and treatment enhancement without pharmacological side effects (Montgomery et al., 2002; Ogez et al., 2024; Rosendahl et al., 2023; Valentine et al., 2019). Preliminary evidence suggests hypnosis can improve attentional control and reduce fatigue in neurological populations (Gilbert et al., 2006; Jensen et al., 2025).

However, research on hypnosis in neurology remains limited, with a need for larger, rigorously controlled studies to confirm its efficacy and understand underlying mechanisms. This feasibility study aims to assess the practicality and acceptability of using hypnosis to treat attentional deficits and fatigue in patients with stroke, TBI, and MS, while also evaluating preliminary efficacy.

A key aspect of this study involves recording electroencephalography (EEG) during both hypnosis and sham-hypnosis sessions. EEG data will provide insight into neural correlates of attentional processing and determine whether hypnosis induces measurable changes in brain activity relative to sham conditions.

ELIGIBILITY:
Inclusion Criteria:

ICD-10 Diagnosis of stroke, TBI or MS Admitted to the inpatient and/or outpatient in the Clinic for Neurology and Neurorehabilitation Age 18 years old or older Understanding the German language Written informed consent

Exclusion Criteria:

Psychiatric disease

Exclusion criteria for the EEG:

Scalp or skin conditions that interfere with EEG electrode placement (e.g. open wounds, infections, severe psoriasis) Implanted medical or neurostimulation devices that interfere with EEG electrode placement (e.g. deep brain stimulators, cochlear implants)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the study design and procedures | From enrollment to the end of treatment at 3 weeks
  The primary objective is to evaluate the feasiblity of conducting the study by assessing the recruitment process, including eligibility and consent rates, determining the participant retention rate troughout the intervention period; conducting baseline assessments, identifying reasons for participants drop-out or non-completion, exploring participant adherence to the intervention protocol and follow-up procedures.

SECONDARY OUTCOMES:
Video-oculography during free visual exploration | Change before and after the intervention over the period of 3 weeks.
  The secondary endpoints are changes in eye movement parameters during free visual exploration (FVE) from pre- to post-intervention, measured by video-oculography (e.g., fixation duration, saccade amplitude, mean gaze positions). Furthermore, between-group differences (hypnosis vs sham-hypnosis) in FVE parameters post-intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Luzerner Kantonsspital, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jensen MP, Barber J, Romano JM, Molton IR, Raichle KA, Osborne TL, Engel JM, Stoelb BL, Kraft GH, Patterson DR. A comparison of self-hypnosis versus progressive muscle relaxation in patients with multiple sclerosis and chronic pain. Int J Clin Exp Hypn. 2009 Apr;57(2):198-221. doi: 10.1080/00207140802665476. PMID 19234967
- [Background] Diamond, S. G., Davis, O. C., Schaechter, J. D., & Howe, R. D. (2006). Hypnosis for rehabilitation after stroke: six case studies. Contemporary hypnosis, 23(4), 173-180.
- [Background] Valentine KE, Milling LS, Clark LJ, Moriarty CL. THE EFFICACY OF HYPNOSIS AS A TREATMENT FOR ANXIETY: A META-ANALYSIS. Int J Clin Exp Hypn. 2019 Jul-Sep;67(3):336-363. doi: 10.1080/00207144.2019.1613863. PMID 31251710
- [Background] Rosendahl J, Alldredge CT, Haddenhorst A. Meta-analytic evidence on the efficacy of hypnosis for mental and somatic health issues: a 20-year perspective. Front Psychol. 2024 Jan 8;14:1330238. doi: 10.3389/fpsyg.2023.1330238. eCollection 2023. PMID 38268815
- [Background] Ogez D, Landry M, Caron-Trahan R, Jusseaux AE, Aubin M, Veronneau J, Fournier V, Godin N, Idrissi M, Rainville P, Richebe P. Make me more comfortable: effects of a hypnosis session on pain perception in chronic pain patients. Front Psychol. 2024 Feb 28;15:1362208. doi: 10.3389/fpsyg.2024.1362208. eCollection 2024. PMID 38481624
- [Background] Montgomery GH, David D, Winkel G, Silverstein JH, Bovbjerg DH. The effectiveness of adjunctive hypnosis with surgical patients: a meta-analysis. Anesth Analg. 2002 Jun;94(6):1639-45, table of contents. doi: 10.1097/00000539-200206000-00052. PMID 12032044
- [Background] Hersche R, Weise A, Michel G, Kesselring J, Bella SD, Barbero M, Kool J. Three-week inpatient energy management education (IEME) for persons with multiple sclerosis-related fatigue: Feasibility of a randomized clinical trial. Mult Scler Relat Disord. 2019 Oct;35:26-33. doi: 10.1016/j.msard.2019.06.034. Epub 2019 Jun 29. PMID 31280074
- [Background] Lefaucheur JP, Aleman A, Baeken C, Benninger DH, Brunelin J, Di Lazzaro V, Filipovic SR, Grefkes C, Hasan A, Hummel FC, Jaaskelainen SK, Langguth B, Leocani L, Londero A, Nardone R, Nguyen JP, Nyffeler T, Oliveira-Maia AJ, Oliviero A, Padberg F, Palm U, Paulus W, Poulet E, Quartarone A, Rachid F, Rektorova I, Rossi S, Sahlsten H, Schecklmann M, Szekely D, Ziemann U. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS): An update (2014-2018). Clin Neurophysiol. 2020 Feb;131(2):474-528. doi: 10.1016/j.clinph.2019.11.002. Epub 2020 Jan 1. PMID 31901449
- [Background] Bode LKG, Sprenger A, Helmchen C, Hauptmann B, Munte TF, Machner B. Combined optokinetic stimulation and cueing-assisted reading therapy to treat hemispatial neglect: A randomized controlled crossover trial. Ann Phys Rehabil Med. 2023 Jun;66(5):101713. doi: 10.1016/j.rehab.2022.101713. Epub 2023 Jan 14. PMID 36645965
- [Background] Rayegani SM, Heidari S, Seyed-Nezhad M, Kiyani N, Moradi-Joo M. Effectiveness of cognitive rehabilitation in comparison with routine rehabilitation methods in patients with multiple sclerosis: A systematic review and meta-analysis. Mult Scler J Exp Transl Clin. 2024 Sep 12;10(3):20552173241272561. doi: 10.1177/20552173241272561. eCollection 2024 Jul-Sep. PMID 39290831
- [Background] Liu-Ambrose T, Falck RS, Dao E, Best JR, Davis JC, Bennett K, Hall PA, Hsiung GR, Middleton LE, Goldsmith CH, Graf P, Eng JJ. Effect of Exercise Training or Complex Mental and Social Activities on Cognitive Function in Adults With Chronic Stroke: A Randomized Clinical Trial. JAMA Netw Open. 2022 Oct 3;5(10):e2236510. doi: 10.1001/jamanetworkopen.2022.36510. PMID 36227593
- [Background] Alashram AR. Computerized cognitive rehabilitation for patients with traumatic brain injury: A systematic review of randomized controlled trials. Appl Neuropsychol Adult. 2024 May 10:1-10. doi: 10.1080/23279095.2024.2350607. Online ahead of print. PMID 38726576
- [Background] Chiaravalloti ND, DeLuca J. Cognitive impairment in multiple sclerosis. Lancet Neurol. 2008 Dec;7(12):1139-51. doi: 10.1016/S1474-4422(08)70259-X. PMID 19007738